CLINICAL TRIAL: NCT03190902
Title: Cognitive Impairment in Pediatric Onset Multiple Sclerosis: Research of Biomarkers Predictive of Cognitive Impairment Progression
Brief Title: Cognitive Impairment in Pediatric Onset Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pietro Iaffaldano (Other)
Responsible Party: Sponsor-Investigator, Pietro Iaffaldano, MD, University of Bari
Organization: University of Bari (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR001
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Pediatric Onset Multiple Sclerosis; ADHD Predominantly Inattentive Type
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Single center, double blind, randomized clinical trial (RCT).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- specific computer training (ST) - POMS (Experimental)
  Interventions: Behavioral: Attention Processing Training program (APT)
- nonspecific computer training (n-ST) - POMS (Active Comparator)
  Interventions: Behavioral: nonspecific computer training (n-ST)
- specific computer training (ST) - ADHD (Experimental)
  Interventions: Behavioral: Attention Processing Training program (APT)
- nonspecific computer training (n-ST) - ADHD (Active Comparator)
  Interventions: Behavioral: nonspecific computer training (n-ST)

INTERVENTIONS:
Behavioral: Attention Processing Training program (APT)
  Arms: specific computer training (ST) - ADHD; specific computer training (ST) - POMS
Behavioral: nonspecific computer training (n-ST)
  Arms: nonspecific computer training (n-ST) - ADHD; nonspecific computer training (n-ST) - POMS

SUMMARY:
Computer-assisted rehabilitation of attention deficits in pediatric Multiple Sclerosis and ADHD patients recruited during the study "Cognitive impairment in Pediatric Onset Multiple Sclerosis: research of biomarkers predictive of cognitive impairment progression".

DETAILED DESCRIPTION:
The presence of cognitive deficits of varied intensity is characteristic of psychiatric disorders of childhood and adolescence such as Attention Deficit Hyperactivity Disorder (ADHD), but also of neurological pathologies such as pediatric onset multiple sclerosis (POMS).

ADHD is one of the most common neurodevelopmental disorders characterized by pervasive patterns of inattention and/or impulsivity/hyperactivity and a range of cognitive dysfunctions that often persist into adulthood.

POMS represent 5-10% of total MS population. Cognitive dysfunction is one of the most remarkable features of MS, and, particularly in POMS, the percentage of patients with at least a mild cognitive deficit ranges from 30 to 80%. The most affected cognitive domains in POMS are complex attention, information processing speed, executive functions, verbal and visual memory, reasoning and problem solving.

The functional consequences of cognitive impairment can be particularly striking in children and adolescents since they occur during formative years in the academic career and may affect their social activities. Cognitive training, during the developmental age, when brain plasticity is at the highest expression, can induce a strengthening of the key brain networks implicated in POMS and ADHD. To date the efficacy of specific cognitive rehabilitation interventions has never been evaluated by a randomized controlled trials (RCTS) in POMS. Conversely, in the last years, several RCTs assessed the efficacy of cognitive training as a potential non-drug alternative treatment for ADHD disorder.Most of the cognitive trainings focused on the working memory or attention dysfunctions. Preliminary evidence suggests that cognitive remediation might be at least partially effective in the ADHD treatment. It is argued that cognitive training can reduce ADHD symptoms and improve functioning by targeting neuropsychological deficits thought to mediate ADHD pathophysiology.

During the study project "Cognitive impairment in Pediatric Onset Multiple Sclerosis: research of biomarkers predictive of cognitive impairment progression", which is aimed to assess clinical, radiological and biological markers in pediatric subjects, POMS and ADHD patients will be recruited to assess the efficacy of a home-based computerized program for retraining attention dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* POMS diagnosed according to the most recent diagnostic criteria;
* age <18 years;
* Expanded Disability Status Scale (EDSS) score ≤5.5;
* impairment on at least 2/4 attention tests defined as scores <1.5 standard deviation (SD) of normative values;
* ADHD patients with the subtype inattention;
* ADHD diagnosis performed according the DSM-5 criteria and the NIMH Collaborative Multisite Multimodal Treatment Study of Children With Attention- Deficit/Hyperactivity Disorder (MTA) - Swanson, Nolan, and Pelham IV Rating Scale (MTA-SNAP-IV), Conner's Parent Rating Scale Revised (CPRS-R), Conner's Teacher Rating Scale Revised (CTRS-R), Child Behavior Checklist (CBCL), Kiddie Schedule for Affective Disorder and Schizophrenia (K-SADS);
* age <18 years;
* impairment on at least 2/4 attention tests defined as scores <1.5 standard deviation (SD) of normative values;

Exclusion Criteria:

* severe cognitive impairment (performance ≤2.0 SD of normative values);
* severe visual loss (unable to read Times New Roman font 16 with the best correction);
* major psychiatric illness;
* alcohol or substance abuse;
* education <5 years;
* previous cognitive rehabilitation training;
* ongoing relapse or steroid treatment during the 30 days preceding enrollment;
* ADHD subtype hyperactivity;
* previously exposure or treatment with any psychotropic drug.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-09-15; Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
to evaluate the effect of the cognitive training on neuropsychological performances. | 3 months
  A global score, defined Cognitive Impairment Index (CII), allowing the evaluation of changes in cognitive performances independently by the number of cognitive tests failed at the neuropsychological evaluation, will be obtained using the mean and SD from the normative values for each test.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simone M, Viterbo RG, Margari L, Iaffaldano P. Computer-assisted rehabilitation of attention in pediatric multiple sclerosis and ADHD patients: a pilot trial. BMC Neurol. 2018 Jun 8;18(1):82. doi: 10.1186/s12883-018-1087-3. PMID 29884144